CLINICAL TRIAL: NCT04361084
Title: To Identify if Mixed Reality Can Produce a Realistic and Adaptable Community Environment for Simulation Compared to Traditional Simulation Techniques.
Brief Title: Community Simulation Utilising Mixed Reality (MR)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Torbay and South Devon NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 264392
Record Dates: First submitted 2020-04-07; First posted 2020-04-24 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Education
Keywords: training; staff; community care

STUDY DESIGN:
Intervention Model Description: This feasibility study involves staff within the host Trust. Staff booking into the training will select available dates. These dates have been randomly assigned (not visible on booking to participants) to do traditional or virtual reality simulation training. Only on attending the actual training day will participants find out which training allocation they will undertake.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional training (Active Comparator): Participants will undertake the Community simulation using traditional methods, physical items to recreate the community environment. Training will be in pairs and will play the role of their own profession when undertaking simulated scenarios. Medium to low fidelity traditional simulation techniques involving scenarios played out using actors as (standardised patients) to participants. Following a briefing, the participants will be asked a series of questions prior to the simulation to establish their profession, age and level of previous training achieved so this can be compared against the results and are anonymous. They will also complete their pre-questionnaire which will anonymous. Afterwards participants undertake a post-questionnaire and then asked if they wish to take part in a semi-structured interview.
  Interventions: Other: traditional simulated training
- mixed reality simulation training (Experimental): Participants will undertake a mixed reality (MR) simulation training session set in two home situations; involving immersive virtual reality equipment. Participants will be asked a series of questions prior to the simulation to establish their profession, age and level of previous training achieved so this can be compared against the results. The participants will then undertake the simulation watched via live camera by the simulation technician, simulation fellow and a community specialist. Participants will undertake a post simulation questionnaire and then asked if they wish to take part in a semi-structured interview (optional).
  Interventions: Other: mixed reality simulation

INTERVENTIONS:
Other: traditional simulated training — traditional simulation using actors as standardised patients playing out scenarios plus pre and post questionnaires and semi structured interviews
  Arms: traditional training
Other: mixed reality simulation — using immersive technologies to create a virtual reality simulated training scenario's plus pre an post questionnaires and semi structured interview's
  Arms: mixed reality simulation training

SUMMARY:
The scope of this project is to identify if mixed reality (MR) can support simulating the complexities of differing community environments compared to traditional physical structure simulated environments. Concurrent with this, the aim is to establish if mixed reality can produce a safe learning and reflective environment for community staff to develop their skills. This could potentially improve patient outcome and support healthcare teams to deliver safe effective care. Evidence suggests that simulation based learning improves confidence; although there is limited research available that combines simulation based learning and mixed reality. As mixed reality could provide high fidelity simulations, it is an area which requires much needed research.

DETAILED DESCRIPTION:
The scope of this project is to identify if mixed reality (MR) can support simulating the complexities of differing community environments compared to traditional physical structure simulated environments. Concurrent with this, the aim is to establish if mixed reality can produce a safe learning and reflective environment for community staff to develop their skills. This could potentially improve patient outcome and support healthcare teams to deliver safe effective care. Simulation is a technique for practice and learning to replace and amplify real experiences with guided ones, and are often immersive in nature. Simulation is a safe, learning environment, that encourages participants to reflect on the situation. Mixed reality is the merging of real and virtual worlds to produce new environment and visualisation where physical and digital objects can co-exist and interact in real time.

For sustainability of the health and social care sector, the long term aim is to facilitate people's healthcare needs in the community. Such increased community services will require staff with holistic skills to work as independent practitioners. Simulation in the acute setting is currently provided by the simulation team in the Trust's dedicated simulation suite, and through in-situ simulations within individual departments. The scenarios for these simulations can be created due to the repetitive and clinical nature of the environments required. Since becoming an integrated care organisation, the need to provide simulation based learning to all staff, including those who are out in community settings has arisen. In order to create a realistic learning environment for community based staff, there is a need to recreate an individual's home, accounting for all of the different environments the investigator's patients live in, such as a small residence with tight spaces, differing levels of cleanliness and the addition of pets, which is very difficult using traditional simulation methods. The need to develop an innovative way of delivering community based simulation is therefore important, to allow all staff access to valuable simulation based learning while providing a safe and supportive environment to practice both technical and non-technical skills.

The investigator proposes to run two simulations per week resulting in undertaking a total of 34 simulations. One of these will be using traditional methods of simulation, and the other will be using mixed reality. Using traditional methods, physical items will be used to recreate the community environment. It can be costly, time consuming and difficult to achieve the desired environment. Mixed reality provides the option of quickly immersing participants into different environments,allowing participants to experience all of the features. This makes it a very useful to method to compare to traditional methods of simulation, as the outcomes could be potentially be more realistic. The investigator will use questionnaires to get feedback from participants, both before, and after they have taken part in the simulation. This feedback will be used to determine if participants feel more confident and competent from traditional methods of simulation or mixed reality based simulation. It will also assess which environment they feel creates a more realistic environment to learn in. Qualitative data will be collected by those participants who choose to take part in a semi-structured interview. Alongside collecting data from participants the simulation technicians will also be asked via a face to face approach to attend a semi-structured interview regarding the feasibility and adaptable of both simulations. This is voluntary. As although participants feedback is important it is also essential that the technician feedback is included as they will be the ones that have to assist with running the simulations. The semi-structured interviews will be undertaken similar to participants semi-structured interviews, with written consent forms, recording of interview and confidentiality. However the questions will be different. They will be given a participant information sheet when they are approached. Evidence suggests that simulation based learning improves confidence; although there is limited research available that combines simulation based learning and mixed reality. As mixed reality could provide high fidelity simulations, it is an area which requires much needed research.

ELIGIBILITY:
Inclusion Criteria:

* Participants need to be full or part time healthcare staff that work within the community setting, patients own homes.

  * These participants can be registered or non-registered staff but needs to be clinical members of staff
  * Staff will be from various professions, including nurses, occupational therapists, physiotherapists, assistant practitioners and support workers. Relying on volunteers, the study is unlikely to have an even representation of all professions, especially bearing in mind numbers of staff within each profession (proportionately more healthcare support workers than specialist therapist).
  * Participants need to be employed, whether full time/part time or on the bank by Torbay and South Devon to be able to participate in this study.
  * As this is only for staff employed by the local trust, this will mean no one under the age of 18 will be included in this study and those staff who are over the age of 80 will also be excluded, as the Trust doesn't employ clinical healthcare professions outside of these age limits.
  * Only healthcare professionals who have given implied consent will be included.

Exclusion Criteria:

* Any individuals who do not work with patients or services users within a community setting (patient's own homes or residential/nursing homes). This will mean non-clinical staff members will be excluded.

  * Participants under the age of 18 and above 80 years old.
  * Participants who are unable to provide informed consent.
  * Participants who have one of the following health conditions will be excluded: Conjunctivitis, Pregnant (5 months+), Corneal Ulcers, Ear infections/ear disease, Corneal Infections, Influenza, "Dry Eye", Head Cold, Iritis, Respiratory Ailments, Cataracts or Glaucoma, Cochlear Implants or other Inner Ear/Vestibular-Related Conditions (e.g.Labyrinthitis). Also anyone that is under the influence of alcohol or drugs on the simulation day. This is due to the unknown research of MR with participants who have medical conditions that could be affected.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate participant confidence following simulated scenario training | 1 year
  Any difference in participants level of learning and confidence following traditional classroom based simulation of clinical community scenarios using actors compared with simulation of scenarios using mixed reality (virtual reality) technology. Assessment using semi structured interviews (N.B no measurement scales involved)

SECONDARY OUTCOMES:
is mixed reality more adaptable and realistic compared to traditional physical (classroom) based simulation environments | 1 year
  Assessment using semi structured interviews (N.B no measurement scales involved)

IPD SHARING:
Plan to Share IPD: No